CLINICAL TRIAL: NCT04297696
Title: Investigation of Effectiveness of Therapeutic Exercises on Target Joint Functions and Gait in Hemophilic Arthropathic Patients.
Brief Title: The Effects of Exercises on Gait in Hemophilic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Volkan Deniz, PT, Director, Cukurova University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 89/55
Record Dates: First submitted 2020-02-29; First posted 2020-03-05 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Hemophilic Arthropathy
Keywords: hemophilia; exercise; gait kinematic
MeSH Terms: conditions — Hemophilia A; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): therapeutic exercises
  Interventions: Other: Therapeutic exercises
- control group (No Intervention)

INTERVENTIONS:
Other: Therapeutic exercises — A program including warm-up period and neuromuscular exercises is applied progressively in two phases.
  Arms: exercise group

SUMMARY:
Arthropathy characterized by synovitis, cartilage degeneration, subchondral and interosseous cysts occur due to hemorrhage in hemophilia. This situation causes to chronic pain, decreasing in range of motion, muscle strength, proprioception. Disorders in these parameters are the main causes of gait dysfunction. The aim of this study is to investigate the effects of therapeutic exercises on target joint functions and gait kinematics, and to determine possible complications related to exercise in hemophilic patients.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed as Hemophilia A or Hemophilia B
* To be over 18 years old
* To have hemophilic arthropathy in at least one joint
* Undergoing prophylaxis or factor VIII-IX replacement therapy

Exclusion Criteria:

* Having another congenital coagulopathy, such as Von Willebrand syndrome
* To be unable to walk due to hemophilic arthropathy
* Having another musculoskeletal problem
* Individuals with inhibitors against Factor VIII-IX

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Haemophilia Joint Health Score | Baseline, Change from baseline HJHS at 2 months, Change from baseline HJHS at 6 months
  Haemophilia Joint Health Score (HJHS) will be applied to evaluate the joint functions of hemophilic individuals. HJHS is a sensitive and valid test used to determine the severity of clinical symptoms that result from hemarthrosis. This comprises an assessment of joints with regards to swelling, muscle atrophy, crepitus, range of motion, joint pain, strength, and global gait. The score for each joint is summed to obtain a total score ranging from 0 to 124, where no joint damage is indicated by a score of 0.
Range of Motion Analysis with Kinovea Software | Baseline, Change from baseline range of motion during gait at 2 months, Change from baseline range of motion during gait at 6 months.
  Range of motion (ROM) analysis during gait will be done by analyzing video images with computer software "Kinovea". Kinovea is a free software used by sports and healthcare professionals to analyze video images during physical activity. Furthermore, it is a sensitive method that can be used to evaluate the range of motion of the lower limb joints during gait. ROM analysis of the ankle and knee joints will be done with Kinovea in the heel strike-midstance-toe off and mid-swing phases.

SECONDARY OUTCOMES:
Haemophilia Quality of Life Questionnaire for Adults | Baseline, Change from baseline 6min-WT at 2 months, Change from baseline Quality of life at 6 months
  The Haem-A-QoL questionnaire including 10 sections and 46 questions was used to evaluate the changes in the Quality of life of PwH; low scores indicate high QoL
Six Minutes Walking Test | Baseline, Change from baseline 6min-WT at 2 months, Change from baseline 6min-WT at 6 months
  Six-Minutes Walking Test (6min-WT) will be applied to determine the effects of therapeutic exercises on the aerobic capacity of hemophilic individuals. This test is a valid and reliable method for determining aerobic capacity in patients with neuromuscular problems. High walking distance indicates high aerobic capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Nevin Atalay Güzel, Prof Dr, Study Director — Gazi University
Locations (1):
- Cukurova University Gym, Adana, Turkey (Türkiye)